CLINICAL TRIAL: NCT04487912
Title: Dynamics and Tracer Distribution of Tilmanocept Using Combined Subareolar and Peritumoral Injection Technique for Scintigraphic Sentinel Lymph Node Detection in Early Stage Breast Cancer
Brief Title: Dynamics and Tracer Distribution of Tilmanocept in Early Stage Breast Cancer
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient patient inclusion
Sponsor: University Hospital, Ghent (Other)
Collaborators: Norgine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: AGO/2019/003
Record Dates: First submitted 2020-07-22; First posted 2020-07-27 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2020-06

CONDITIONS: Breast Cancer; Sentinel Lymph Node
MeSH Terms: conditions — Breast Neoplasms | interventions — technetium Tc 99m nanocolloid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Injection of 99m-Tc Tilmanocept (Active Comparator)
  Interventions: Drug: Tilmanocept
- Injection of 99m-Tc Nanocolloid (Active Comparator)
  Interventions: Drug: Nanocolloid

INTERVENTIONS:
Drug: Tilmanocept — Combined peri-areolar and peri-tumoral injection of 99m-Tc Tilmanocept
  Arms: Injection of 99m-Tc Tilmanocept
Drug: Nanocolloid — Combined peri-areolar and peri-tumoral injection of 99m-Tc Nanocolloid
  Other Names: Nanoscint
  Arms: Injection of 99m-Tc Nanocolloid

SUMMARY:
A sentinel node procedure is recommended for patients with early stages of breast cancer to exclude metastases to local lymph nodes. This procedure is done with a "tracer" which is injected near to the tumor and drains to these nearby lymph nodes. The first draining lymph node(s) are called "sentinel" node(s). These sentinel nodes are excised by the surgeon for microscopic investigation using a detection probe. This study aims to further document the distribution and dynamics of a recently approved new tracer called Tilmanocept and comparing it with the standard used tracer (nanocolloid) to determine whether there is a significant difference between both products (which are both approved for clinical use in this scenario in the European Union). This will be done by randomly assigning patients between injection of Tilmanocept or Nanocolloid and making scans on multiple (3) time points.

ELIGIBILITY:
Inclusion Criteria:

* Early stage breast cancer (T1, T2)
* Clinically node negative (no enlarged axillary lymph nodes)

Exclusion Criteria:

* Prior surgery in same breast
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Time to identification of first lymph node | 0-30 minutes
  Time to identification of first lymph node on the dynamic acquisition during the first 30 minutes post-injection
Lymph node count to background ratio 4 hours post-injection | 4 hours post-injection
  Number of identified lymph nodes and count-to-background ratio in these identified lymph nodes obtained by SPECT/CT 4 hours post-injection
Lymph node count to background ratio 24 hours post-injection | 20 to 24 hours post-injection
  Number of identified lymph nodes and count-to-background ratio in these identified lymph nodes obtained by SPECT/CT 24 hours post-injection
Injection site count to background ratio 4 hours post-injection | 4 hours post-injection
  Count-to-background ratio in the radionuclide injection sites obtained by SPECT/CT 4 hours post-injection
Injection site count to background ratio 24 hours post-injection | 20 to 24 hours post-injection
  Count-to-background ratio in the radionuclide injection sites obtained by SPECT/CT 24 hours post-injection

CONTACTS AND LOCATIONS:
Locations (1):
- university hospital, Ghent, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giammarile F, Alazraki N, Aarsvold JN, Audisio RA, Glass E, Grant SF, Kunikowska J, Leidenius M, Moncayo VM, Uren RF, Oyen WJ, Valdes Olmos RA, Vidal Sicart S. The EANM and SNMMI practice guideline for lymphoscintigraphy and sentinel node localization in breast cancer. Eur J Nucl Med Mol Imaging. 2013 Dec;40(12):1932-47. doi: 10.1007/s00259-013-2544-2. Epub 2013 Oct 2. PMID 24085499
- [Background] Unkart JT, Hosseini A, Wallace AM. Tc-99m tilmanocept versus Tc-99m sulfur colloid in breast cancer sentinel lymph node identification: Results from a randomized, blinded clinical trial. J Surg Oncol. 2017 Dec;116(7):819-823. doi: 10.1002/jso.24735. Epub 2017 Jul 10. PMID 28695567
- [Background] Unkart JT, Proudfoot J, Wallace AM. Outcomes of "one-day" vs "two-day" injection protocols using Tc-99m tilmanocept for sentinel lymph node biopsy in breast cancer. Breast J. 2018 Jul;24(4):526-530. doi: 10.1111/tbj.13002. Epub 2018 Mar 2. PMID 29498443